CLINICAL TRIAL: NCT01567839
Title: Anesthetic Efficacy of 4% Articaine With 1:100,000 Epinephrine, 4% Prilocaine With 1:200,000 Epinephrine, and 4% Lidocaine With 1:100,000 Epinephrine as a Primary Buccal Infiltration in the Mandibular First Molar.
Brief Title: Testing the Anesthetic Effectiveness of Three Different Dental Local Anesthetics Injected Next to a Lower First Molar
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, John Nusstein, Associate Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 4% dental local anesthetics
Record Dates: First submitted 2012-03-28; First posted 2012-03-30 (Estimated); Results first posted 2014-01-01 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-11

CONDITIONS: Anesthetic Effectiveness
Keywords: degree of pulpal anesthesia obtained; primary infiltration in the lower first molar

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 4% Lidocaine (Experimental): 1.8 mL of 4% lidocaine with 1:100,000 epinephrine
  Interventions: Procedure: Mandibular buccal Infiltration injection
- 4% Articaine (Experimental): 1.8 mL of 4% articaine with 1:100,000 epinephrine
  Interventions: Procedure: Mandibular buccal Infiltration injection
- 4% Prilocaine (Experimental): 1.8 mL of 4% prilocaine with 1:200,000 epinephrine
  Interventions: Procedure: Mandibular buccal Infiltration injection

INTERVENTIONS:
Procedure: Mandibular buccal Infiltration injection

SUMMARY:
Infiltration (injecting next to the tooth) injections are common in dentistry and a number of studies have shown that articaine anesthetic, when injected next to the tooth as a supplemental injection, works very well following a typical inferior alveolar (lower jaw) nerve block. No study has compared 4% articaine with 1:100,000 epinephrine, 4% prilocaine with 1:200,000 epinephrine, and 4% lidocaine with 1:100,000 epinephrine in mandibular (lower jaw) infiltration injections of the first molar. The purpose of this prospective, randomized, double-blind, crossover study is to compare the degree of anesthesia obtained from the three solutions as a primary infiltration injection next to the mandibular first molar. The investigators also will record the pain of injection and postoperative pain.

DETAILED DESCRIPTION:
Using a crossover design, 60 adult subjects will receive three injections consisting of a primary mandibular first molar infiltration of 1.8 mL of 4% articaine with 1:100,000 epinephrine, 1.8 mL of 4% prilocaine with 1:200,000 epinephrine, and 1.8 mL of 4% lidocaine with 1:100,000 epinephrine in three separate appointments spaced at least one week apart. With the crossover design, 180 infiltrations will be given for the first molar and each subject will serve as his or her own control. Ninety infiltrations will be administered on the mandibular left side and ninety administered on the mandibular right side. The order of the three injections will be assigned randomly and the dentist and subject will be blinded about which anesthetic the subject is given. The anesthetics used in this study are not experimental. An electric pulp tester will be used to test the lower back teeth (molars and premolars) for anesthesia in 3-minute time intervals for a total of 60 minutes. The pain of injection and postoperative pain will be recorded in a survey. The data will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 65 years.
* in good health (ASA classification II or lower).
* able to provide informed consent.

Exclusion Criteria:

* allergy to articaine, lidocaine or prilocaine.
* history of significant medical problems (ASA classification III or greater).
* depression (taking tri-cyclic antidepressant medications to control).
* have taken CNS depressants (including alcohol or any analgesic medications) within the last 48 hours prior to testing.
* lactating or pregnant.
* inability to give informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-05; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University College of Dentistry, Postle Hall, Columbus, Ohio, United States

REFERENCES:
- [Background] Kanaa MD, Whitworth JM, Corbett IP, Meechan JG. Articaine buccal infiltration enhances the effectiveness of lidocaine inferior alveolar nerve block. Int Endod J. 2009 Mar;42(3):238-46. doi: 10.1111/j.1365-2591.2008.01507.x. PMID 19228214
- [Background] Kanaa MD, Whitworth JM, Corbett IP, Meechan JG. Articaine and lidocaine mandibular buccal infiltration anesthesia: a prospective randomized double-blind cross-over study. J Endod. 2006 Apr;32(4):296-8. doi: 10.1016/j.joen.2005.09.016. Epub 2006 Feb 17. PMID 16554198
- [Background] Robertson D, Nusstein J, Reader A, Beck M, McCartney M. The anesthetic efficacy of articaine in buccal infiltration of mandibular posterior teeth. J Am Dent Assoc. 2007 Aug;138(8):1104-12. doi: 10.14219/jada.archive.2007.0324. PMID 17670879
- [Background] Haase A, Reader A, Nusstein J, Beck M, Drum M. Comparing anesthetic efficacy of articaine versus lidocaine as a supplemental buccal infiltration of the mandibular first molar after an inferior alveolar nerve block. J Am Dent Assoc. 2008 Sep;139(9):1228-35. doi: 10.14219/jada.archive.2008.0338. PMID 18762633
- [Background] Corbett IP, Kanaa MD, Whitworth JM, Meechan JG. Articaine infiltration for anesthesia of mandibular first molars. J Endod. 2008 May;34(5):514-8. doi: 10.1016/j.joen.2008.02.042. PMID 18436027
- [Background] Abdulwahab M, Boynes S, Moore P, Seifikar S, Al-Jazzaf A, Alshuraidah A, Zovko J, Close J. The efficacy of six local anesthetic formulations used for posterior mandibular buccal infiltration anesthesia. J Am Dent Assoc. 2009 Aug;140(8):1018-24. doi: 10.14219/jada.archive.2009.0313. PMID 19654255

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment at the College of Dentistry between May 2012 and December 2012.
Pre-assignment Details: No exclusions. All subjects enrolled were utilized and assigned.
Groups:
- Subjects Receiving Injections: All subjects received each of the three anesthetic injections.
Period: Overall Study
Arm/Group | Subjects Receiving Injections
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: No difference.
Arm/Group | Subjects Receiving Injections
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25.8 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 30
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Successful Pulpal Anesthesia.
Description: Two consecutive 80/80 readings (no patient response) during 60 minutes of testing with an electric pulp tester.
Time Frame: 60 minutes
Measure: Number; unit: participants
Arm/Group | 4% Articaine With 1:100,000 Epinephrine | 4% Lidocaine With 1:100,000 Epinephrine | 4% Prilocaine With 1:200,000 Epinephrine
Number analyzed (Participants) | 60 | 60 | 60
participants
  Second Molar | 37 | 27 | 22
  First Molar | 33 | 20 | 19
  Second Premolar | 32 | 21 | 17
  First Premolar | 29 | 24 | 18

ADVERSE EVENTS:
Arm/Group | 4% Articaine With 1:100,000 Epinephrine | 4% Lidocaine With 1:100,000 Epinephrine | 4% Prilocaine With 1:200,000 Epinephrine
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60

LIMITATIONS AND CAVEATS:
No adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes